CLINICAL TRIAL: NCT00005425
Title: Statistical Analysis of Vlagtwedde-Vlaardingen Data Set
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4343; R03HL049460 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2001-04

CONDITIONS: Asthma; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To determine the effects in early adulthood of asthma, increased bronchial responsiveness, markers of allergy and smoking on pulmonary function level and the effects of these same risk factors on subsequent decline in pulmonary function, because these early adult factors presumably profoundly influence the risk for chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The questions studied included whether the above named risk factors reduced the maximally attained level of pulmonary function in early adulthood, foreshortened the postulated stability of level of pulmonary function between age 18 and 35 and/or unfavorably affected subsequent decline in level of pulmonary function. FEV1/h2, VC/h2 and FEV1/IVC were studied, using graphic smooth techniques and regression analyses techniques on both cross-sectional and longitudinal datasets. In addition, the investigators tested the hypothesis stating that early adult symptoms of asthma, increased bronchial responsiveness, markers of allergy influenced who became a smoker, influenced the amount smoked and/or influenced who stopped smoking relatively early in adult life, using logistic regression analyses and survival analyses.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1995-02 (Actual)

REFERENCES:
- [Background] Shimada M, Matsumata T, Itasaka H, Shirabe K, Taketomi A, Sugimachi K. The prediction of portal pressure: a multivariate analysis of clinical data and intraoperative portal pressure. Surg Today. 1994;24(4):309-12. doi: 10.1007/BF02348558. PMID 8038504
- [Background] Xu X, Weiss ST, Dockery DW, Schouten JP, Rijcken B. Comparing FEV1 in adults in two community-based studies. Chest. 1995 Sep;108(3):656-62. doi: 10.1378/chest.108.3.656. PMID 7656612
- [Background] Rijcken B, Schouten JP, Xu X, Rosner B, Weiss ST. Airway hyperresponsiveness to histamine associated with accelerated decline in FEV1. Am J Respir Crit Care Med. 1995 May;151(5):1377-82. doi: 10.1164/ajrccm.151.5.7735588.
- [Background] Xu X, Laird N, Dockery DW, Schouten JP, Rijcken B, Weiss ST. Age, period, and cohort effects on pulmonary function in a 24-year longitudinal study. Am J Epidemiol. 1995 Mar 15;141(6):554-66. doi: 10.1093/oxfordjournals.aje.a117471. PMID 7900723